CLINICAL TRIAL: NCT02929147
Title: Comparison of Efficacy and Safety of the Postoperative Analgesia Methods for Supratentorial Craniotomy by Integrated Pulmonary Index (IPI)
Brief Title: Comparison of Efficacy and Safety of the Postoperative Analgesia Methods
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Özlem Korkmaz Dilmen, MD, DESA, Associate Prof. in Anesthesiology, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Istanbul U
Record Dates: First submitted 2016-10-06; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Supratentorial Neoplasms
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Morphine; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Morphine 1 mg (Experimental): In the Group 1 the PCA will set to administer a bolus dose of 1 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours.
  Interventions: Drug: Morphine
- Morphine 0.5 (Experimental): In the Group 2 the PCA set to administer a bolus dose of 0.5 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours
  Interventions: Drug: Morphine
- Dexketoprofen & Placebo (Active Comparator): The Group 3 will take 50 mg dexketoprofen in the recovery room. Intra venous injections of dexketoprofen will repeat every 8 hours.
  Interventions: Drug: Dexketoprofen; Drug: Placebo

INTERVENTIONS:
Drug: Morphine — In the Group 1 the PCA will set to administer a bolus dose of 1 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours. In the Group 2 the PCA set to administer a bolus dose of 0.5 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours.
  Arms: Morphine 0.5; Morphine 1 mg
Drug: Dexketoprofen — The Group 3 will take 50 mg dexketoprofen in the recovery room. Intra venous injections of dexketoprofen will repeat every 8 hours.
  Other Names: Arveles
  Arms: Dexketoprofen & Placebo
Drug: Placebo — In the Group 3 the PCA will contain placebo.
  Other Names: SF
  Arms: Dexketoprofen & Placebo

SUMMARY:
An optimal analgesic therapy is very important for postoperative recovery. In recent years, several studies showed that the prevalence of the moderate to severe pain after craniotomy ranged from 69 to 87% of patients. In a previous study, the investigators showed that the use of morphine based patient controlled analgesia prevented moderate to severe postoperative pain in patients undergoing supratentorial craniotomy. Morphine related side effects such as sedation, miosis, respiratory depression, nausea and vomiting produce a general reluctance for their use in neurosurgery. Therefore, all patients were closely observed to detect opioid related side effects in the intensive care unit for 24 hours following surgery in the previous study. The Integrated Pulmonary Index (IPI) is a new tool that calculates respiratory and hemodynamic parameters noninvasively. In the present study the investigators will use different doses of morphine based PCA and the IPI system to determine more effective and safer morphine dose for postoperative analgesia following supratentorial craniotomy.

DETAILED DESCRIPTION:
An optimal analgesic therapy is very important for postoperative recovery. In recent years, several studies showed that the prevalence of the moderate to severe pain after craniotomy ranged from 69 to 87% of patients. In a previous study, the investigators showed that the use of morphine based patient controlled analgesia prevented moderate to severe postoperative pain in patients undergoing supratentorial craniotomy. Morphine related side effects such as sedation, miosis, respiratory depression, nausea and vomiting produce a general reluctance for their use in neurosurgery. Therefore, all patients were closely observed to detect opioid related side effects in the intensive care unit for 24 hours following surgery in the previous study. The Integrated Pulmonary Index (IPI) is a new tool that calculates respiratory and hemodynamic parameters noninvasively. In the present study the investigators will use different doses of morphine based PCA and the IPI system to determine more effective and safer morphine dose for postoperative analgesia following supratentorial craniotomy.

90 patients will randomize in 3 groups following supratentorial craniotomy. All patients will previously instruct on the PCA pumps (Abbott Provider, Chicago, USA) and visual analogue scale (VAS) from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. All patients will use PCA for 24 hours following supratentorial craniotomy. In the Group 1 the PCA will set to administer a bolus dose of 1 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours. In the Group 2 the PCA set to administer a bolus dose of 0.5 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours. In the Group 3 the PCA will contain placebo. The Group 3 will take 50 mg dexketoprofen in the recovery room. Intra venous injections of dexketoprofen will repeat every 8 hours. If the VAS skore more than 4 the Group 3 patients will take 1 g paracetamol every 6 hours.

All patients will observe by the Integrated Pulmonary Index (IPI). It is a new device that provides to recognise in a patients respiratory status. This software tool is a single index value ranging from 1 to 10 based on 4 physiological parameters: end tidal carbon dioxide, respiratory rate, oxygen saturation, pulse rate. Patients will asses at 10th minute, 1, 2, 6, 12, and 24 hours postoperatively. Sedation will evaluate according to Ramsay score. VAS scores, total morphine consumption, Ramsay score, blood pressure, heart rate and respiratory rate, the IPI score will record at each time pain will evaluate. Postoperative side effects, including rash, pruritus, nausea and vomiting will record at the same intervals and defined by a scale with 0 = absent or 1 = present. Moreover the lowest IPI score, the apnea count (longer than 30 seconds) and the count of the desaturation events will record in the postoperative 24 hours.

The 3 Groups will compare with respect to VAS scores, morphine consumption, IPI scores, the apnea count, the desaturation events and morphine related side effects during the 24 hours following supratentorial craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of supratentorial neoplasms

Exclusion Criteria:

* Neurological disorders hindering the communication, aphasia, Glasgow Coma Score (GCS) less than 15, drug or alcohol addiction, chronic pain, raised intracranial pressure, allergies to any of the drugs used in this study, hepatic or renal dysfunction, peptic ulcer disease, dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Integrated Pulmonary Index (IPI) | Change from Beseline IPI values in postoperative first 24 hours.(at 10th minute, 1, 2, 6, 12, and 24 hours post dose)

SECONDARY OUTCOMES:
Pain intensity measured by Visual Analog Score | Change from Beseline Pain Intensity in postoperative first 24 hours(at 10th minute, 1, 2, 6, 12, and 24 hours post dose)
Sedation level measured by Ramsay score | Change from Beseline Sedation Level in postoperative first 24 hours(at 10th minute, 1, 2, 6, 12, and 24 hours post dose)
Cumulative Morphine consumption | Change from Baseline in 1postoperative first 24 hours(at 10th minute, 1, 2, 6, 12, and 24 hours post dose)

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Korkmaz Dilmen, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Ozlem Korkmaz Dilmen, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dilmen OK, Akcil EF, Tunali Y, Karabulut ES, Bahar M, Altindas F, Vehid H, Yentur E. Postoperative analgesia for supratentorial craniotomy. Clin Neurol Neurosurg. 2016 Jul;146:90-5. doi: 10.1016/j.clineuro.2016.04.026. Epub 2016 May 4. PMID 27164511
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Garah J, Adiv OE, Rosen I, Shaoul R. The value of Integrated Pulmonary Index (IPI) monitoring during endoscopies in children. J Clin Monit Comput. 2015 Dec;29(6):773-8. doi: 10.1007/s10877-015-9665-z. Epub 2015 Feb 11. PMID 25666393
- [Derived] Akcil EF, Korkmaz Dilmen O, Ertem Vehid H, Yentur E, Tunali Y. The role of "Integrated Pulmonary Index" monitoring during morphine-based intravenous patient-controlled analgesia administration following supratentorial craniotomies: a prospective, randomized, double-blind controlled study. Curr Med Res Opin. 2018 Nov;34(11):2009-2014. doi: 10.1080/03007995.2018.1501352. Epub 2018 Aug 5. PMID 30010438